CLINICAL TRIAL: NCT06045559
Title: Effects of Sevoflurane, Desflurane or Propofol Anesthesia on High-Dose Rocuronium in Laparoscopic Cholecystectomy Operations
Brief Title: Effects of Anesthetics on High-Dose Rocuronium
Status: Recruiting | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Selim Turhanoglu, Professor Dr., Mustafa Kemal University
Other Study IDs: 2022/38
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Neuromuscular Blockade; Anesthetic Agents
Keywords: inhalational anesthetics; Neuromuscular Blockade; rocuronium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- S(Sevoflurane): Anesthesia induction for all patients will be performed with 2 mg/kg propofol and 2 µg/kg fentanyl. Following loss of eyelash reflex, 1.2 mg/kg rocuronium will be administered intravenously to all patients. Anesthesia will be maintained with sevoflurane, with a BIS value between 40-50 and a minimal alveolar concentration (MAC) value between 1-1.5.
- D(Desflurane): Anesthesia induction for all patients will be performed with 2 mg/kg propofol and 2 µg/kg fentanyl. Following loss of eyelash reflex, 1.2 mg/kg rocuronium will be administered intravenously to all patients. Anesthesia will be maintained with desflurane, with a BIS value between 40-50 and a MAC value between 1-1.5.
- P(Propofol): Anesthesia induction for all patients will be performed with 2 mg/kg propofol and 2 µg/kg fentanyl. Following loss of eyelash reflex, 1.2 mg/kg rocuronium will be administered intravenously to all patients. Propofol was administered intravenously at a rate of 6-12 mg/kg/min to maintain anesthesia, keeping the BIS value between 40-50.

SUMMARY:
This study evaluates the effects of three different anesthetics on high dose rocuronium in laparoscopic cholecystectomy cases. Patients were randomly assigned to one of the propofol, desflurane, or sevoflurane groups. Train of four (TOF) and bispectral index (BIS) monitoring were used during surgery in all groups.Patients were followed until TOF and post tetanic count (PTC) values reached 1 and the time was recorded.The effect of three anesthetic drugs used on the duration of the muscle relaxant drug was investigated.

DETAILED DESCRIPTION:
In recent years, studies have been published showing that by applying deep neuromuscular block during laparoscopic cholecystectomy, intraabdominal pressure can be reduced without compromising the surgical conditions, thus complications such as postoperative nausea and vomiting (PONV) and pain can be reduced.

The results we obtained in our previous study showed that deep neuromuscular block achieved with a high dose of 1.2 mg/kg rocuronium allowed the operation to be performed with lower intra-abdominal pressure values, shortened the operation time, reduced PONV and pain in laparoscopic cholecystectomy cases. The most important factor affecting the depth of neuromuscular block is the dose of the neuromuscular agent. However, anesthetic agents can also affect the depth of neuromuscular blockade. The effects of muscle relaxants are enhanced when administered together with inhalation anesthetics.Propofol and sevoflurane are widely used in the maintenance of anesthesia. Unlike propofol, sevoflurane enhances the effects of some neuromuscular blocking drugs, including rocuronium.

Our primary aim in this study is to evaluate the effects of sevoflurane, desflurane, or propofol, which are commonly used in anesthesia maintenance, on the duration of neuromuscular block caused by 1.2 mg/kg rocuronium, which is the dose we routinely use in anesthesia induction, in laparoscopic cholecystectomy cases. Secondary aims are to investigate its effects on intraabdominal pressures and surgical conditions, and to determine whether it reduces postoperative pain and PONV, as well as extubation and recovery times.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) Ⅰ-Ⅲ patients
* between the ages of 18-65

Exclusion Criteria:

* Being under 18 of age or over 65
* disapproval of the informed consent
* rocuronium allergy
* sugammadex allergy
* pregnancy
* lactation
* hepatic or renal dysfunction
* obesity (BMI≥35kg/m2)
* Previous abdominal surgery
* long-term use of NSAIs
* neuromuscular disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 65 who applied to our hospital for laparoscopic cholecystectomy surgery from October 2023 to June 2024.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
Duration of neuromuscular block with rocuronium. | 15 seconds for TOF rates, 8 minutes for PTC values
  TOF rates will be measured every 15 seconds and PTC values will be measured every 8 minutes. Additionally, the times of TOF 0 and PTC 0 responses and TOF1 and PTC 1 responses will be recorded.

SECONDARY OUTCOMES:
intra-abdominal pressure | 5 minutes
  Effect of deep neuromuscular block on intra-abdominal pressure
surgical conditions | It will be evaluated once at the end of the surgery based on the surgeon's satisfaction.
  Effect of deep neuromuscular block on surgical conditions
postoperative pain | 2nd, 24th and 72nd hours after surgery
  Effect of deep neuromuscular block on postoperative pain
postoperative nausea and vomiting | postoperative 4th, 12th and 24th hours
  The effect of deep neuromuscular blockade on postoperative nausea and vomiting will be evaluated.
Length of extubation process | 15sc
  Time from discontinuation of maintenance anesthesia to extubation.
Lenght of recovery process | 1 mınute
  Time from extubation to modified Aldrete score of 9.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Turhanoglu, MD, Principal Investigator — Mustafa Kemal University; Serhat Hakkoymaz, MD, Study Director — Mustafa Kemal University; Menekşe Okşar, MD, Study Director — Mustafa Kemal University; Muhyittin Temiz, MD, Study Director — Mustafa Kemal University; Emre Dirican, Study Director — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Antakya, Hatay, Turkey (Türkiye)